CLINICAL TRIAL: NCT05430204
Title: Continuous Glucose Monitoring for Screening for Diabetes in Pregnancy:A Comparative Effectiveness Randomized Control Trial (PRECISE)
Brief Title: Continuous Glucose Monitoring for Screening for Diabetes in Pregnancy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: DexCom, Inc. (Industry)
Responsible Party: Principal Investigator, Michal Fishel Bartal, Assistant Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: HSC-MS-22-0153
Record Dates: First submitted 2022-06-14; First posted 2022-06-24 (Actual); Results first posted 2025-12-04 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Gestational Diabetes
MeSH Terms: conditions — Diabetes, Gestational

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- one-hour Glucose tolerance test (GCT) (Active Comparator)
  Interventions: Device: Group 1: one-hour GCT
- CGM screening (Experimental)
  Interventions: Device: Group 2: CGM placement

INTERVENTIONS:
Device: Group 1: one-hour GCT — Group I will be comprised of one-hour 50g glucose challenge participants for diagnosis of GDM..Diagnosis will be based on 1-hour glucose challenge test results: 1-hour result ≤ 130 mg/dL, the participant will have passed the challenge test. 1-hour result ≥ 130 mg/dL will complete a three-hour 100g glucose tolerance test. If two out of three values are elevated per Carpenter Coustan criteria , the participant will be diagnosed with GDM and treated according to the standard of care. This group will also receive the CGM.CGM data will not be observed until completion of study and will not be available to provider. Participants will return transmitter at follow up visit after completion of 7 days.Group I will receive routine prenatal care follow-up depending upon one-hour glucose results as written above.
  Arms: one-hour Glucose tolerance test (GCT)
Device: Group 2: CGM placement — CGM will consist of using the Dexcom G6 Pro device. The device will be placed on the abdomen or the arm.The Dexcom G6/G7 Pro App will be downloaded on the patient's phone. A patient profile will be created on the Dexcom Clarity portal .The patient will receive an email to link their portal to the clinic's portal.The patient will receive a message through Epic electronic medical records to remove the CGM 10 days after placement.The device will be reviewed by the Diabetes team 48 hours after CGM is removed. The recommended range for glucose during pregnancy is defined as 63-140 mg/dL .The time above range has been defined as ≥ 140 mg/dL, greater than 10% of total CGM placement time. The following criteria will currently be used to diagnose gestational diabetes in the CGM group:
  * Time above range (≥140 mg/dL) ≥ 10% of the time while using CGM or
  * Average glucose≥130 mg/dL or
  * Any glucose value ≥200 mg/dL
  Arms: CGM screening

SUMMARY:
The purpose of this study is to evaluate whether Continuous glucose monitoring (CGM) for diagnosis of gestational diabetes mellitus (GDM) improves maternal and neonatal outcomes related to GDM and to evaluate whether CGM for GDM diagnosis reduces the health system costs for mother-infant dyads compared to usual care

ELIGIBILITY:
Inclusion Criteria:

* 24-30 weeks gestation undergoing GDM screening

Exclusion Criteria:

* Known diagnosis of Type I and II DM
* History of bariatric surgery
* Major fetal anomalies
* Unwilling to use CGM for GDM screening
* Incarcerated subjects
* History of allergic reaction to any of CGM metals or adhesives in contact with the skin

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1628 (Actual)
Dates: Start 2023-03-07 (Actual); Primary Completion 2024-08-02 (Actual); Study Completion 2024-09-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michal Fishel Bartal, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fishel Bartal M, Ashby Cornthwaite J, Ghafir D, Ward C, Nazeer SA, Blackwell SC, Pedroza C, Chauhan SP, Sibai BM. Continuous glucose monitoring in individuals undergoing gestational diabetes screening. Am J Obstet Gynecol. 2023 Oct;229(4):441.e1-441.e14. doi: 10.1016/j.ajog.2023.04.021. Epub 2023 Apr 23. PMID 37088275

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 1,628 individuals (814 mother-infant dyads) were enrolled. Each mother was enrolled during pregnancy, prior to the birth of her infant. Following delivery, data collection continued for both mother and infant as part of the same dyad.
Period: Overall Study
Arm/Group | CGM screening | one-hour Glucose tolerance test (GCT)
Started | 405 (A total of 405 Infant-mother dyads were in the CGM screening arm. Each mother was enrolled during pregnancy, prior to the birth of her infant. Following delivery, data collection continued for both mother and infant as part of the same dyad.) | 409 (A total of 409 Infant-mother dyads were in the one-hour Glucose tolerance test (GCT) arm. Each mother was enrolled during pregnancy, prior to the birth of her infant. Following delivery, data collection continued for both mother and infant as part of the same dyad.)
Completed | 388 (A total of 388 Infant-mother dyads completed the study in the CGM screening arm. Each mother was enrolled during pregnancy, prior to the birth of her infant. Following delivery, data collection continued for both mother and infant as part of the same dyad.) | 392 (A total of 392 Infant-mother dyads completed the study in the one-hour Glucose tolerance test (GCT). Each mother was enrolled during pregnancy, prior to the birth of her infant. Following delivery, data collection continued for both mother and infant as part of the same dyad.)
Not Completed | 17 | 17

BASELINE CHARACTERISTICS:
Population: Baseline Characteristics were not collected for infants.
Groups:
- Total: Total of all reporting groups
Arm/Group | CGM Screening | One-hour Glucose Tolerance Test (GCT) | Total
Number analyzed (Participants) | 405 | 409 | 814
Age, Continuous [Mean (Standard Deviation); unit: years] | 29 (5.9) | 29 (6.4) | 29 (6.15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 405 | 409 | 814
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Non-Hispanic White | 77 | 59 | 136
  Non-Hispanic Black | 144 | 145 | 289
  Hispanic | 117 | 142 | 259
  Unknown | 67 | 63 | 130
Region of Enrollment [Number; unit: participants]
  United States | 405 | 409 | 814
Number of maternal participants on government assisted insurance [Count of Participants; unit: Participants] | 263 | 269 | 532
Number of maternal participants with Nulliparous [Count of Participants; unit: Participants] — Nulliparous means never given birth before.
  Participants | 124 | 136 | 260
Number of maternal participants with body mass index (BMI) greater than 30 at first prenatal visit [Count of Participants; unit: Participants] | 215 | 245 | 460
Number of maternal participants with body mass index (BMI) greater than 40 [Count of Participants; unit: Participants] | 70 | 73 | 143
Number of maternal participants with chronic hypertension [Count of Participants; unit: Participants] | 36 | 38 | 74
Number of maternal participants with family history of diabetes mellitus [Count of Participants; unit: Participants] | 180 | 168 | 348
Number of maternal participants with Gestational diabetes in previous pregnancy [Count of Participants; unit: Participants] | 24 | 29 | 53
Gestational age at randomization [Mean (Standard Deviation); unit: weeks] | 26.0 (1.6) | 25.8 (1.5) | 25.89 (1.55)
Number of maternal participants with Thyroid disease [Count of Participants; unit: Participants] | 22 | 16 | 38
Number of maternal participants with tobacco use during pregnancy [Count of Participants; unit: Participants] | 8 | 3 | 11
Number of maternal participants with Alcohol use during pregnancy [Count of Participants; unit: Participants] | 4 | 5 | 9
Number of maternal participants with Substance use during pregnancy [Count of Participants; unit: Participants] | 8 | 7 | 15

OUTCOME MEASURES:

1. Primary Outcome: Number of Neonates That Show Composite Adverse Neonatal Outcome
Description: Composite adverse neonatal outcome include one or more of the following:
  * Large for Gestational Age(LGA) is described as weight over 90th percentile of the expected value according to gestational age (using the nomogram by Duryea EL et al)
  * Shoulder Dystocia is defined as the need for any extra maneuvers, other than gentle downward traction of the fetal head to deliver the fetal body after the fetal head has been delivered
  * Birth injury: skull, clavicular, humerus fracture, or brachial plexus injury
  * Neonatal hypoglycemia: less than 40 mg/dL in the first 24 hours of life and less than 50 mg/dL after or requiring medical therapy
  * Respiratory distress is described as the need for at least 4 hours of respiratory support with supplemental oxygen, continuous positive airway pressure, or ventilation at the first 24 hours of life
  * Fetal or neonatal death (within 28 days of birth)
Time Frame: From birth to about 28 days of life.
Measure: Count of Participants; unit: Participants
Arm/Group | CGM screening | one-hour Glucose tolerance test (GCT)
Number analyzed (Participants) | 388 | 392
Participants | 130 | 114

2. Primary Outcome: Number of Neonates That Show Adverse Neonatal Outcome of Large for Gestational Age(LGA)
Description: LGA is described as weight over 90th percentile of the expected value according to gestational age (using the nomogram by Duryea EL et al)
Time Frame: at time of birth
Measure: Count of Participants; unit: Participants
Arm/Group | CGM screening | one-hour Glucose tolerance test (GCT)
Number analyzed (Participants) | 388 | 392
Participants | 32 | 29

3. Primary Outcome: Number of Neonates That Show Adverse Neonatal Outcome of Shoulder Dystocia
Description: Shoulder dystocia is defined as the need for any extra maneuvers, other than gentle downward traction of the fetal head to deliver the fetal body after the fetal head has been delivered
Time Frame: at time of birth
Measure: Count of Participants; unit: Participants
Arm/Group | CGM screening | one-hour Glucose tolerance test (GCT)
Number analyzed (Participants) | 388 | 392
Participants | 5 | 3

4. Primary Outcome: Number of Neonates That Show Adverse Neonatal Outcome of Birth Injury
Description: Birth injury: skull, clavicular, humerus fracture, or brachial plexus injury
Time Frame: at time of birth
Measure: Count of Participants; unit: Participants
Arm/Group | CGM screening | one-hour Glucose tolerance test (GCT)
Number analyzed (Participants) | 388 | 392
Participants | 1 | 0

5. Primary Outcome: Number of Neonates That Show Adverse Neonatal Outcome of Neonatal Hypoglycemia
Description: Neonatal hypoglycemia: less than 40 mg/dL in the first 24 hours of life and less than 50 mg/dL after or requiring medical therapy
Time Frame: from birth to discharge (about 3-15 days)
Measure: Count of Participants; unit: Participants
Arm/Group | CGM screening | one-hour Glucose tolerance test (GCT)
Number analyzed (Participants) | 388 | 392
Participants | 87 | 68

6. Primary Outcome: Number of Neonates That Show Adverse Neonatal Outcome of Respiratory Distress
Description: Respiratory distress is described as the need for at least 4 hours of respiratory support with supplemental oxygen, continuous positive airway pressure, or ventilation at the first 24 hours of life
Time Frame: from birth to discharge (about 3-15 days)
Measure: Count of Participants; unit: Participants
Arm/Group | CGM screening | one-hour Glucose tolerance test (GCT)
Number analyzed (Participants) | 388 | 392
Participants | 45 | 47

7. Primary Outcome: Number of Fetal or Neonatal Deaths
Time Frame: within 28 days of birth
Measure: Count of Participants; unit: Participants
Arm/Group | CGM screening | one-hour Glucose tolerance test (GCT)
Number analyzed (Participants) | 388 | 392
Participants | 2 | 2

8. Secondary Outcome: Feasibility as Assessed by the Number of Participants Who Complete the CGM Diagnostic Testing
Time Frame: From enrollment to 6 weeks post partum, on average 21 weeks
Population: Data for this outcome measure were only collected for participants in the GCM screening arm.
Measure: Count of Participants; unit: Participants
Arm/Group | CGM screening | one-hour Glucose tolerance test (GCT)
Number analyzed (Participants) | 405 | 0
Participants | 388 |

9. Secondary Outcome: Number of Women That Use Diabetic Medication During Pregnancy
Description: diabetic medication is described as any glycemic control agent
Time Frame: From enrollment to 6 weeks post partum, on average 21 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | CGM screening | one-hour Glucose tolerance test (GCT)
Number analyzed (Participants) | 388 | 392
Participants
  Metformin | 7 | 9
  Insulin | 21 | 8

10. Secondary Outcome: Number of Women That Show Polyhydramnios During Pregnancy Not Related to Known Fetal Anomaly
Time Frame: From enrollment to delivery
Measure: Count of Participants; unit: Participants
Arm/Group | CGM screening | one-hour Glucose tolerance test (GCT)
Number analyzed (Participants) | 388 | 392
Participants | 63 | 67

11. Secondary Outcome: Number of Women That Have Preterm Birth
Description: Pre term birth is described as delivery less than 37 weeks of gestation
Time Frame: at time of birth
Measure: Count of Participants; unit: Participants
Arm/Group | CGM screening | one-hour Glucose tolerance test (GCT)
Number analyzed (Participants) | 388 | 392
Participants | 68 | 65

12. Secondary Outcome: Number of Women That Undergo Induced Labor
Time Frame: at time of birth
Measure: Count of Participants; unit: Participants
Arm/Group | CGM screening | one-hour Glucose tolerance test (GCT)
Number analyzed (Participants) | 388 | 392
Participants | 194 | 207

13. Secondary Outcome: Number of Women That Experience Pregnancy Induced Hypertension
Time Frame: From enrollment to 6 weeks post partum, on average 21 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | CGM screening | one-hour Glucose tolerance test (GCT)
Number analyzed (Participants) | 388 | 392
Participants | 63 | 71

14. Secondary Outcome: Number of Women That Experience Eclampsia: Seizures
Time Frame: From enrollment to 6 weeks post partum, on average 21 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | CGM screening | one-hour Glucose tolerance test (GCT)
Number analyzed (Participants) | 388 | 392
Participants | 0 | 0

15. Secondary Outcome: Number of Women Admitted Due to Poor Glucose Control
Time Frame: From enrollment up to delivery
Measure: Count of Participants; unit: Participants
Arm/Group | CGM screening | one-hour Glucose tolerance test (GCT)
Number analyzed (Participants) | 388 | 392
Participants | 1 | 0

16. Secondary Outcome: Number of Women With Primary Cesarean Section
Time Frame: at time of birth
Measure: Count of Participants; unit: Participants
Arm/Group | CGM screening | one-hour Glucose tolerance test (GCT)
Number analyzed (Participants) | 388 | 392
Participants | 67 | 73

17. Secondary Outcome: Number of Women With Postpartum Hemorrhage: Defined as Greater Then 1000ml
Time Frame: From enrollment to 6 weeks post partum, on average 21 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | CGM screening | one-hour Glucose tolerance test (GCT)
Number analyzed (Participants) | 388 | 392
Participants | 17 | 18

18. Secondary Outcome: Number of Women With Endometritis
Time Frame: From enrollment to 6 weeks post partum, on average 21 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | CGM screening | one-hour Glucose tolerance test (GCT)
Number analyzed (Participants) | 388 | 392
Participants | 6 | 4

19. Secondary Outcome: Number of Women With Wound Complications
Time Frame: From enrollment to 6 weeks post partum, on average 21 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | CGM screening | one-hour Glucose tolerance test (GCT)
Number analyzed (Participants) | 388 | 392
Participants | 1 | 1

20. Secondary Outcome: Number of Women With Diagnosis of Type 2 Diabetes During Postpartum
Time Frame: birth to 6 weeks postpartum
Measure: Count of Participants; unit: Participants
Arm/Group | CGM screening | one-hour Glucose tolerance test (GCT)
Number analyzed (Participants) | 388 | 392
Participants | 2 | 1

21. Secondary Outcome: Number of Neonates With Apgar Score Less Than 7
Description: The Apgar score is determined by evaluating the newborn baby on each of five criteria (appearance, pulse, grimace, activity, respiration) on a scale from zero to two, then summing the five values obtained. The total score ranges from zero to 10. A higher score indicates a better outcome.
Time Frame: 5 minutes after birth
Measure: Count of Participants; unit: Participants
Arm/Group | CGM screening | one-hour Glucose tolerance test (GCT)
Number analyzed (Participants) | 388 | 392
Participants | 17 | 18

22. Secondary Outcome: Number of Neonates That Are Admitted to the Neonatal Intensive Care Unit (NICU)
Time Frame: birth to time of discharge from NICU (about 15 days)
Measure: Count of Participants; unit: Participants
Arm/Group | CGM screening | one-hour Glucose tolerance test (GCT)
Number analyzed (Participants) | 388 | 392
Participants | 69 | 74

23. Secondary Outcome: NICU Length of Stay
Time Frame: birth to time of discharge from NICU (about 15 days)
Measure: Mean (Inter-Quartile Range); unit: hours
Arm/Group | CGM screening | one-hour Glucose tolerance test (GCT)
Number analyzed (Participants) | 388 | 392
hours | 100 [48 to 303.5] | 123.5 [48.0 to 360.0]

24. Secondary Outcome: Number of Neonates With Hyperbilirubinemia Requiring Phototherapy
Time Frame: birth to discharge (about 3-15 days)
Measure: Count of Participants; unit: Participants
Arm/Group | CGM screening | one-hour Glucose tolerance test (GCT)
Number analyzed (Participants) | 388 | 392
Participants | 32 | 33

25. Secondary Outcome: Number of Neonates With Need for Intravenous or Oral Administration Glucose Therapy
Time Frame: birth to discharge (about 3-15 days)
Measure: Count of Participants; unit: Participants
Arm/Group | CGM screening | one-hour Glucose tolerance test (GCT)
Number analyzed (Participants) | 388 | 392
Participants | 75 | 60

26. Secondary Outcome: Number of Neonates That Are Small for Gestational Age
Description: Small for gestational age, defined as a weight below 10th percentile of the expected value according to gestational age (using the nomogram published by Duryea EL et al)
Time Frame: at time of birth
Measure: Count of Participants; unit: Participants
Arm/Group | CGM screening | one-hour Glucose tolerance test (GCT)
Number analyzed (Participants) | 388 | 392
Participants | 41 | 39

27. Secondary Outcome: Number of Participants Who Breastfed Their Babies
Time Frame: from birth to 6 weeks postpartum
Measure: Count of Participants; unit: Participants
Arm/Group | CGM screening | one-hour Glucose tolerance test (GCT)
Number analyzed (Participants) | 388 | 392
Participants | 121 | 141

28. Secondary Outcome: Number of Participants Who Formula Fed Their Babies
Time Frame: from birth to 6 weeks postpartum
Measure: Count of Participants; unit: Participants
Arm/Group | CGM screening | one-hour Glucose tolerance test (GCT)
Number analyzed (Participants) | 388 | 392
Participants | 75 | 74

29. Secondary Outcome: Maximum Bilirubin Level - Neonates
Time Frame: birth to discharge (about 3 -15 days)
Population: The study team decided that this outcome measure was not going to be collected therefore, the laboratory assays were not performed and no data were collected for this outcome. This outcome will not be collected in the future. The Study Protocol was not amended to reflect this collective team decision
Arm/Group | CGM screening | one-hour Glucose tolerance test (GCT)
Number analyzed (Participants) | 0 | 0

30. Secondary Outcome: Cord Arterial pH
Time Frame: at time of birth
Measure: Mean (Inter-Quartile Range); unit: pH
Arm/Group | CGM screening | one-hour Glucose tolerance test (GCT)
Number analyzed (Participants) | 388 | 392
pH | 7.2 [7.2 to 7.3] | 7.2 [7.2 to 7.3]

31. Secondary Outcome: Number of Neonates With Polycythemia
Time Frame: birth to discharge (about 3 -15 days)
Measure: Count of Participants; unit: Participants
Arm/Group | CGM screening | one-hour Glucose tolerance test (GCT)
Number analyzed (Participants) | 388 | 392
Participants | 32 | 33

32. Secondary Outcome: Number of Women That Experience Preeclampsia With Severe Features
Time Frame: From enrollment to 6 weeks post partum, on average 21 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | CGM screening | one-hour Glucose tolerance test (GCT)
Number analyzed (Participants) | 388 | 392
Participants | 24 | 26

33. Secondary Outcome: Number of Women That Experience Super Imposed Preeclampsia
Time Frame: From enrollment to 6 weeks post partum, on average 21 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | CGM screening | one-hour Glucose tolerance test (GCT)
Number analyzed (Participants) | 388 | 392
Participants | 15 | 17

34. Secondary Outcome: Number of Women With Need for Blood Transfusion
Time Frame: From enrollment to 6 weeks post partum, on average 21 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | CGM screening | one-hour Glucose tolerance test (GCT)
Number analyzed (Participants) | 388 | 392
Participants | 22 | 24

35. Secondary Outcome: Number of Participants With Ultrasound Diagnosis of Estimated Fetal Weight >90%Ile in the Third Trimester
Time Frame: Third trimester (≥28 weeks gestation through delivery)
Measure: Count of Participants; unit: Participants
Arm/Group | CGM screening | one-hour Glucose tolerance test (GCT)
Number analyzed (Participants) | 388 | 392
Participants | 5 | 4

36. Secondary Outcome: Number of Women That Experience HELLP Syndrome
Description: HELLP syndrome: a group of symptoms in pregnant women characterized by hemolysis (H), elevated liver enzymes (EL), and/or low platelet (LP) count, assessed according to ACOG guidelines.
Time Frame: From enrollment to 6 weeks post partum, on average 21 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | CGM screening | one-hour Glucose tolerance test (GCT)
Number analyzed (Participants) | 388 | 392
Participants | 0 | 0

37. Secondary Outcome: Cord Venous pH
Time Frame: at time of birth
Population: Data were not collected or analyzed for Cord Venous pH. The study team determined that collection of cord venous pH was not required based on academic evidence that a different marker, arterial pH, is a reliable marker. This outcome will not be collected in the future. The Study Protocol was not amended to reflect this collective team decision. Please see outcome #30 for data on arterial pH.
Arm/Group | CGM screening | one-hour Glucose tolerance test (GCT)
Number analyzed (Participants) | 0 | 0

38. Secondary Outcome: Total Health System Costs for Mothers and Infants
Time Frame: From enrollment to 6 weeks post partum, on average 21 weeks
Population: Data were not collected or analyzed for this outcome because there was no standardized cost or charging across participants therefore there was no data to collect or analyze for any participants. This outcome will not be collected in the future. The Study Protocol was not amended to reflect this collective team decision
Arm/Group | CGM screening | one-hour Glucose tolerance test (GCT)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Mothers were assessed from enrollment up to 6 weeks post delivery, on average 21 weeks. Infants were assessed from birth up to 6 weeks post delivery, on average 6 weeks.
Groups:
- CGM screening: Infants; CGM screening: Mothers: Group 2: CGM placement: CGM will consist of using the Dexcom G6 Pro device. The device will be placed on the abdomen or the arm.The Dexcom G6/G7 Pro App will be downloaded on the patient's phone. A patient profile will be created on the Dexcom Clarity portal .The patient will receive an email to link their portal to the clinic's portal.The patient will receive a message through Epic electronic medical records to remove the CGM 10 days after placement.The device will be reviewed by the Diabetes team 48 hours after CGM is removed. The recommended range for glucose during pregnancy is defined as 63-140 mg/dL .The time above range has been defined as ≥ 140 mg/dL, greater than 10% of total CGM placement time. The following criteria will currently be used to diagnose gestational diabetes in the CGM group:
  * Time above range (≥140 mg/dL) ≥ 10% of the time while using CGM or
  * Average glucose≥130 mg/dL or
  * Any glucose value ≥200 mg/dL
- one-hour Glucose tolerance test (GCT): Infants; one-hour Glucose tolerance test (GCT): Mothers: Group 1: one-hour GCT: Group I will be comprised of one-hour 50g glucose challenge participants for diagnosis of GDM..Diagnosis will be based on 1-hour glucose challenge test results: 1-hour result ≤ 130 mg/dL, the participant will have passed the challenge test. 1-hour result ≥ 130 mg/dL will complete a three-hour 100g glucose tolerance test. If two out of three values are elevated per Carpenter Coustan criteria , the participant will be diagnosed with GDM and treated according to the standard of care. This group will also receive the CGM.CGM data will not be observed until completion of study and will not be available to provider. Participants will return transmitter at follow up visit after completion of 7 days.Group I will receive routine prenatal care follow-up depending upon one-hour glucose results as written above.
Arm/Group | CGM screening: Infants | one-hour Glucose tolerance test (GCT): Infants | CGM screening: Mothers | one-hour Glucose tolerance test (GCT): Mothers
All-Cause Mortality (participants affected / at risk) | 2/405 | 2/409 | 0/405 | 0/409
Serious Adverse Events (participants affected / at risk) | 0/405 | 0/409 | 0/405 | 0/409
Other Adverse Events (participants affected / at risk) | 0/405 | 0/409 | 0/405 | 0/409

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-07-05): https://cdn.clinicaltrials.gov/large-docs/04/NCT05430204/Prot_SAP_000.pdf